CLINICAL TRIAL: NCT02170051
Title: Improving Negative Symptoms of Psychosis In Real-world Environments
Acronym: INSPIRE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Diego (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Elizabeth Twamley, Professor of Psychiatry, University of California, San Diego
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 130424; 1R34MH101250 (NIH)
Record Dates: First submitted 2014-06-18; First posted 2014-06-23 (Estimated); Results first posted 2020-11-27 (Actual); Last update posted 2021-05-19 (Actual); Status verified 2021-04

CONDITIONS: Schizophrenia
Keywords: negative symptoms; cognition; functioning; defeatist attitudes; psychosocial treatment
MeSH Terms: conditions — Schizophrenia

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- CBSST-CCT (Experimental): Cognitive Behavioral Social Skills Training-Compensatory Cognitive Training
  Interventions: Behavioral: CBSST-CCT
- Goal-focused supportive contact (Active Comparator): Goal-focused supportive contact
  Interventions: Behavioral: Goal focused supportive contact

INTERVENTIONS:
Behavioral: CBSST-CCT
  Other Names: Cognitive Behavioral Social Skills Training-Compensatory Cognitive Training
  Arms: CBSST-CCT
Behavioral: Goal focused supportive contact
  Arms: Goal-focused supportive contact

SUMMARY:
This study will compare Cognitive Behavioral Social Skills Training-Compensatory Cognitive Training (CBSST-CCT) to a goal-focused supportive contact group to see which intervention better improves symptoms and functioning in people with schizophrenia.

ELIGIBILITY:
Inclusion Criteria:

MUST BE A RESIDENT OF BROADWAY HOME, SAN DIEGO, OR A SERVICE USER OF THE MEETING PLACE, ARETA CROWELL, OR PROJECT ENABLE.

1. Voluntary informed consent to participate
2. Age 18 to 65
3. DSM-IV diagnosis of schizophrenia or schizoaffective disorder based on MINI/SCID
4. Moderate-to-severe negative symptoms on the Clinical Assessment Interview for Negative Symptoms (CAINS total score >19)
5. ≥ 6th grade reading level on the Wide Range Achievement Test-4 Reading subtest (needed for reading treatment manual)
6. Stable on medications; no changes within 3 months prior to enrollment

Exclusion Criteria:

1. Prior CBT, SST, or CCT in the past 5 years
2. Severe positive symptoms on the Positive and Negative Syndrome Scale (PANSS Delusions, Disorganization, Hallucinations, or Suspiciousness >5)
3. Severe depression on the Calgary Depression Scale for Schizophrenia (CDSS >8)
4. Ocular damage/disease/surgery/medications that affect pupil dilation
5. DSM-IV alcohol or substance dependence diagnosis in past 6 months based on the MINI or SCID
6. Level of care required interferes with outpatient therapy (e.g., hospitalized; severe medical illness) .

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2014-07-01 (Actual); Primary Completion 2018-09-03 (Actual); Study Completion 2018-09-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth Twamley, PhD, Principal Investigator — UCSD; Eric Granholm, PhD, Principal Investigator — UCSD
Locations (1):
- UCSD, La Jolla, California, United States

REFERENCES:
- [Derived] Granholm E, Twamley EW, Mahmood Z, Keller AV, Lykins HC, Parrish EM, Thomas ML, Perivoliotis D, Holden JL. Integrated Cognitive-Behavioral Social Skills Training and Compensatory Cognitive Training for Negative Symptoms of Psychosis: Effects in a Pilot Randomized Controlled Trial. Schizophr Bull. 2022 Mar 1;48(2):359-370. doi: 10.1093/schbul/sbab126. PMID 34665853

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 2 participants received the wrong diagnosis, and were withdrawn from the study; 7 participants had a CAINS score of ≤19, and were excluded from the study
Groups:
- CBSST-CCT: Cognitive Behavioral Social Skills Training-Compensatory Cognitive Training
  CBSST-CCT
- Goal-focused Supportive Contact: Goal-focused supportive contact
  Goal focused supportive contact
Period: Overall Study
Arm/Group | CBSST-CCT | Goal-focused Supportive Contact
Started | 26 | 29
Tested at Mid-point | 13 | 18
Tested at Post-treatment | 15 | 16
Completed (Tested at 6-month follow-up) | 15 | 16
Not Completed | 11 | 13
Not completed — Withdrawal by Subject | 10 | 10
Not completed — Lost to Follow-up | 1 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | CBSST-CCT | Goal-focused Supportive Contact | Total
Number analyzed (Participants) | 26 | 29 | 55
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 26 | 28 | 54
  >=65 years | 0 | 1 | 1
Age, Continuous [Mean (Standard Deviation); unit: years] | 47.7 (11.4) | 53.2 (7.4) | 50.6 (9.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 13 | 22
  Male | 17 | 16 | 33
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 8 | 10 | 18
  Not Hispanic or Latino | 18 | 19 | 37
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 2 | 0 | 2
  Black or African American | 11 | 4 | 15
  White | 12 | 24 | 36
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 26 | 29 | 55

OUTCOME MEASURES:

1. Primary Outcome: Clinical Assessment Interview for Negative Symptoms (CAINS)
Description: Change in negative symptom severity at 12.5 weeks. Scores range from 0-52; higher values indicate greater severity.
Time Frame: baseline, 12.5 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | CBSST-CCT | Goal-focused Supportive Contact
Number analyzed (Participants) | 15 | 17
score on a scale | .0667 (4.02611) | -.0588 (5.85737)

2. Secondary Outcome: MATRICS Consensus Cognitive Battery (MCCB)
Description: Change in cognitive performance in several domains at 12.5 weeks. Scores range from 0-80; higher scores indicate better performance.
Time Frame: baseline, 12.5 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | CBSST-CCT | Goal-focused Supportive Contact
Number analyzed (Participants) | 15 | 17
score on a scale | .8778 (3.40143) | -.0065 (2.87904)

3. Secondary Outcome: UCSD Performance-based Skills Assessment-Brief (UPSA-B)
Description: Change in communication and financial functioning at 12.5 weeks. Scores range from 0-100; higher scores indicate better performance.
Time Frame: baseline, 12.5 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | CBSST-CCT | Goal-focused Supportive Contact
Number analyzed (Participants) | 15 | 17
score on a scale | 3.1667 (13.91000) | 1.3882 (10.42682)

4. Secondary Outcome: Social Skills Performance Assessment (SSPA)
Description: Change in social skills performance at 12.5 weeks. Scores range from 2-10; higher scores indicate better social skills.
Time Frame: baseline, 12.5 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | CBSST-CCT | Goal-focused Supportive Contact
Number analyzed (Participants) | 15 | 17
score on a scale | .1824 (.56812) | .0548 (.43854)

5. Secondary Outcome: Specific Levels of Functioning Scale (SLOF)
Description: Change in self-reported functioning at 12.5 weeks. Scores range from 30-150. Higher score indicates better functioning.
Time Frame: baseline, 12.5 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | CBSST-CCT | Goal-focused Supportive Contact
Number analyzed (Participants) | 15 | 17
score on a scale | .1718 (.38527) | .2498 (.63886)

6. Secondary Outcome: Independent Living Skills Survey (ILSS)
Description: Change in self-reported functioning at 12.5 weeks. Scores range from 0-1; higher score indicates better skills.
Time Frame: baseline, 12.5 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | CBSST-CCT | Goal-focused Supportive Contact
Number analyzed (Participants) | 15 | 15
score on a scale | .0121 (.04379) | -.0078 (.06717)

7. Secondary Outcome: Defeatist Performance Attitudes Scale (DPAS)
Description: Change in defeatist attitudes at 12.5 weeks. Likert Scale 1-7; scores range from 15-105; higher scores indicate a more severe defeatist performance attitude.
Time Frame: baseline, 12.5 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | CBSST-CCT | Goal-focused Supportive Contact
Number analyzed (Participants) | 15 | 17
score on a scale | -3.8667 (11.01860) | 1.1765 (19.38825)

8. Secondary Outcome: Scale for the Assessment of Negative Symptoms (SANS)
Description: Change in negative symptom severity at 12.5 weeks. Scores range from 0-25; higher values indicate greater severity.
Time Frame: baseline, 12.5 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | CBSST-CCT | Goal-focused Supportive Contact
Number analyzed (Participants) | 15 | 17
score on a scale | -.8000 (2.45531) | -.1176 (2.95555)

ADVERSE EVENTS:
Time Frame: 10.5 months
Arm/Group | CBSST-CCT | Goal-focused Supportive Contact
All-Cause Mortality (participants affected / at risk) | 0/26 | 0/29
Serious Adverse Events (participants affected / at risk) | 0/26 | 0/29
Other Adverse Events (participants affected / at risk) | 0/26 | 0/29

LIMITATIONS AND CAVEATS:
High participant dropout rate, leading to a smaller number of subjects analyzed than anticipated.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-10-19): https://cdn.clinicaltrials.gov/large-docs/51/NCT02170051/Prot_SAP_000.pdf